CLINICAL TRIAL: NCT03390842
Title: A Blinded, Placebo-Controlled Extension to Study TRCA-301 to Evaluate the Long-term Safety and Durability of Effect of TRC101 in Subjects With Chronic Kidney Disease and Metabolic Acidosis
Brief Title: Long-term Safety Extension to Study TRCA-301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tricida, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRCA-301E
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Metabolic Acidosis
Keywords: blood bicarbonate, kidney disease
MeSH Terms: conditions — Acidosis; Kidney Diseases | interventions — veverimer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TRC101 (Experimental): Administered once daily (QD) for 40 weeks
  Interventions: Drug: TRC101
- Placebo (Placebo Comparator): Administered once daily (QD) for 40 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRC101 — Oral suspension
  Other Names: Veverimer
  Arms: TRC101
Drug: Placebo — Oral suspension
  Arms: Placebo

SUMMARY:
This study is a 40-week, blinded, placebo-controlled extension of Study TRCA-301 (NCT03317444). Eligible subjects who complete the 12-week treatment period in Study TRCA-301 have the option to participate in this extension study evaluating the long-term safety and durability of effect of TRC101 in subjects with non-dialysis dependent chronic kidney disease and metabolic acidosis. Eligible subjects will be treated with TRC101 or placebo once daily (QD) on an out-patient basis for the subsequent 40 weeks. Subjects will continue to receive the same blinded treatment (TRC101 or placebo) that they received in Study TRCA-301.

ELIGIBILITY:
Key Inclusion Criteria:

* Completed the 12-week treatment period and attended the Week 12 Visit in the parent study TRCA-301.
* Blood bicarbonate level of >= 12 mEq/L at the Week 12 Visit in the parent study TRCA-301.

Key Exclusion Criteria:

* Any level of low blood bicarbonate at the Week 12 Visit that, in the opinion of the Investigator, requires emergency intervention or evaluation for an acute acidotic process.
* Required dialysis for acute kidney injury or worsening CKD during the parent study TRCA-301.
* Planned initiation of renal replacement therapy within 6 months following study entry.
* History or current diagnosis of diabetic gastroparesis, bowel obstruction, swallowing disorders, severe gastrointestinal disorders, inflammatory bowel disease, major gastrointestinal surgery, or active gastric/duodenal ulcers.
* Serum calcium <= 8.0 mg/dL at the Week 10 in the parent study TRCA-301.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Tricida, Inc.
Locations (29):
- United States (7):
  - Investigative Site 55, Phoenix, Arizona
  - Investigative Site 91, Los Angeles, California
  - Investigative Site 59, Hialeah, Florida
  - Investigative Site 93, Hollywood, Florida
  - Investigative Site 92, Lauderdale Lakes, Florida
  - Investigative Site 95, Atlanta, Georgia
  - Investigative Site 52, San Antonio, Texas
- Investigative Site 11, Sofia, Bulgaria
- Georgia (7):
  - Investigative Site 31, Tbilisi
  - Investigative Site 32, Tbilisi
  - Investigative Site 33, Tbilisi
  - Investigative Site 34, Tbilisi
  - Investigative Site 35, Tbilisi
  - Investigative Site 36, Tbilisi
  - Investigative Site 37, Tbilisi
- Hungary (4):
  - Investigative Site 41, Budapest
  - Investigative Site 46, Budapest
  - Investigative Site 49, Hódmezővásárhely
  - Investigative Site 44, Kistarcsa
- Investigative Site 61, Vršac, Serbia
- Slovenia (2):
  - Investigative Site 72, Jesenice
  - Investigative Site 71, Maribor
- Ukraine (7):
  - Investigative Site 81, Kharkiv
  - Investigative Site 83, Kharkiv
  - Investigative Site 87, Kharkiv
  - Investigative Site 88, Kharkiv
  - Investigative Site 84, Kyiv
  - Investigative Site 85, Kyiv
  - Investigative Site 86, Kyiv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wesson DE, Mathur V, Tangri N, Stasiv Y, Parsell D, Li E, Klaerner G, Bushinsky DA. Long-term safety and efficacy of veverimer in patients with metabolic acidosis in chronic kidney disease: a multicentre, randomised, blinded, placebo-controlled, 40-week extension. Lancet. 2019 Aug 3;394(10196):396-406. doi: 10.1016/S0140-6736(19)31388-1. Epub 2019 Jun 24. PMID 31248662
- [Derived] Mathur VS, Wesson DE, Tangri N, Li E, Bushinsky DA. Effects of veverimer on serum bicarbonate and physical function in women with chronic kidney disease and metabolic acidosis: a subgroup analysis from a randomised, controlled trial. BMC Nephrol. 2022 Feb 25;23(1):82. doi: 10.1186/s12882-022-02690-1. PMID 35216581

RESULTS

PARTICIPANT FLOW:
Groups:
- TRC101 Treatment Arm: TRC101 was self-administered orally as an aqueous suspension, QD with food, at approximately the same time each day for 40 weeks. Subjects entered the study on the same blinded TRC101 dose they were receiving in the parent study, TRCA-301, as follows: 0, 3, 6 or 9 g TRC101 QD (0, 1, 2 or 3 packets, respectively). Subjects could have had a blinded dose adjustment using these same doses in accordance with a protocol-specified titration algorithm at each study visit.
- Placebo Treatment Arm: Placebo was self-administered orally as an aqueous suspension, QD with food, at approximately the same time each day for 40 weeks. Subjects entered the study on the same blinded placebo dose they were receiving in the parent study, TRCA-301, as follows: 0, 1, 2 or 3 placebo packets QD. Subjects could have had a blinded dose adjustment using these same doses in accordance with a protocol-specified titration algorithm at each study visit.
Period: Overall Study
Arm/Group | TRC101 Treatment Arm | Placebo Treatment Arm
Started | 114 | 82
Completed | 111 | 74
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRC101 Treatment Arm | Placebo Treatment Arm | Total
Number analyzed (Participants) | 114 | 82 | 196
Age, Categorical [Count of Participants; unit: Participants] — Age (years) was calculated as the number of years between date of birth and date of informed consent in the parent study TRCA-301, expressed as an integer.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 56 | 44 | 100
    >=65 years | 58 | 38 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] — Age (years) was calculated as the number of years between date of birth and date of informed consent in the parent study TRCA-301, expressed as an integer.
  years | 62.9 (12.07) | 61.7 (11.88) | 62.4 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 31 | 77
  Male | 68 | 51 | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 113 | 79 | 192
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
History of Hypertension [Count of Participants; unit: Participants] | 110 | 79 | 189
History of Diabetes Mellitus [Count of Participants; unit: Participants] | 70 | 57 | 127
History of Congestive Heart Failure [Count of Participants; unit: Participants] | 34 | 28 | 62
Baseline eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Baseline eGFR is defined as the average of values of eGFR collected at the Screening 1 Visit, Screening 2 Visit, and Baseline Visit (i.e., Day 1 pre-dose) in the parent study TRCA-301, as measured by the central laboratory, based on serum creatinine values using the CKD-EPI formula.
  mL/min/1.73m^2 | 29.4 (6.41) | 27.9 (5.42) | 28.8 (6.05)
Baseline Bicarbonate [Mean (Standard Deviation); unit: mEq/L] — Baseline Bicarbonate is defined as the average of the values of serum bicarbonate collected at the Screening 1 Visit, Screening 2 Visit, and Baseline Visit (i.e., Day 1 pre-dose) in the parent study TRCA-301, measured onsite using an i-STAT point-of-care device.
  mEq/L | 17.21 (1.429) | 17.13 (1.501) | 17.17 (1.457)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events, Serious Adverse Events, and Adverse Events Leading to Withdrawal.
Description: The incidence of adverse events (AEs), serious adverse events (SAEs) and AEs leading to withdrawal. For incidence of AEs and SAEs, see Adverse Events Section. For incidence of AEs leading to withdrawal, see endpoint values below.
Time Frame: Week 12 Visit in the parent study, TRCA-301, to the Week 54 Visit in the extension study, TRCA-301E.
Population: The TRCA-301E Safety Analysis Set included all subjects who received any amount of study drug (TRC101 or placebo) in Study TRCA-301E.
Measure: Number; unit: percentage of participants
Arm/Group | TRC101 Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 112 | 81
percentage of participants | 0 | 1.2

2. Secondary Outcome: Subjects With Change From Baseline in Serum Bicarbonate of ≥ 4 mEq/L or Serum Bicarbonate Within the Normal Range
Description: Percent of subjects having a change from baseline in serum bicarbonate of at least 4 mEq/L or bicarbonate in the normal range (22 - 29 mEq/L) at the end of treatment (Week 52).
Time Frame: Baseline in the parent study, TRCA-301, to the Week 52 Visit in the extension study, TRCA-301E.
Population: The TRCA-301E Modified Intent-to-Treat (MITT) Analysis Set included all randomized subjects who had both baseline and at least one postbaseline serum bicarbonate value measured using the i-STAT device in the parent study, TRCA-301, and at least one serum bicarbonate value after the Week 12 Visit in Study TRCA-301E.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TRC101 Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 110 | 74
percentage of participants | 62.7 [53.0 to 71.8] | 37.8 [26.8 to 49.9]
Statistical Analysis 1: Comparison: TRC101 Treatment Arm vs Placebo Treatment Arm; % Subjects Who Met Endpoint (≥ 4 mEq/L Change from Baseline Serum Bicarbonate or Serum Bicarbonate in the Normal Range [22 - 29 mEq/L]): TRC101-Placebo; Test type: Superiority; p = 0.0015, Fisher Exact; Difference in % of subjects = 24.9, 95% CI 2-sided [10.2 to 38.7]
Statistical Analysis 2: Comparison: TRC101 Treatment Arm vs Placebo Treatment Arm; % Subjects with ≥ 4mEq/L Change from Baseline in Serum Bicarbonate: TRC101-Placebo; Test type: Superiority; p = 0.0015, Fisher Exact; Treatment difference in % of subjects = 24.4, 95% CI 2-sided [9.7 to 38.2]
Statistical Analysis 3: Comparison: TRC101 Treatment Arm vs Placebo Treatment Arm; % Subjects with Serum Bicarbonate in Normal Range (22 - 29 mEq/L): TRC101-Placebo; Test type: Superiority; p < 0.0001, Fisher Exact; Treatment difference in % of subjects = 30.2, 95% CI 2-sided [15.6 to 43.7]

3. Secondary Outcome: Change From Baseline in Serum Bicarbonate at the End of Treatment
Description: Change from baseline in serum bicarbonate at the end of treatment (Week 52).
Time Frame: Baseline in the parent study, TRCA-301, to the Week 52 Visit in the extension study, TRCA-301E.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | TRC101 Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 114 | 82
mEq/L | 4.70 (0.335) | 2.71 (0.403)
Statistical Analysis 1: Comparison: TRC101 Treatment Arm vs Placebo Treatment Arm; Least Squares Mean Change from Baseline: TRC101-Placebo; Test type: Superiority; p = 0.0002, Mixed-effect repeated measures model; Treatment difference in LS means = 1.99, 95% CI 2-sided [0.96 to 3.03], Standard Error of Mean 0.524 — Standard error presented above is for the LS mean

4. Secondary Outcome: Change From Baseline in the Total Score of the KDQOL-PFD at the End of Treatment
Description: Change from baseline in the total score of the Kidney Disease Quality of Life Physical Function Domain (KDQOL-PFD) at the end of treatment. The KDQOL is a validated, kidney disease-specific measure of health-related quality of life. For study TRCA-301E, and the parent study TRCA-301, the 10-question Item 3 of the KDQOL, also known as the SF-36 Physical Function subscale, was selected to measure physical functioning and is referenced herein as the KDQOL-PFD. The KDQOL-PFD was chosen as a patient-reported outcome measurement to evaluate the effects of TRC101 on daily activities that may be adversely affected by loss of muscle caused by metabolic acidosis. The minimum score for each of the 10 questions is 0 (physical activity highly limited) and the maximum is 100 (physical activity not limited). The total KDQOL-PFD score is calculated by adding the scores for all 10 questions, for a minimum and maximum possible total KDQOL-PFD score of 0 or 100, respectively.
Time Frame: Baseline in the parent study, TRCA-301, to the Week 52 Visit in the extension study, TRCA-301E.
Population: as for outcome 2
Measure: Mean (Standard Error); unit: KDQOL-PFD total score
Arm/Group | TRC101 Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 113 | 78
KDQOL-PFD total score | 11.42 (2.201) | -0.71 (2.268)
Statistical Analysis 1: Comparison: TRC101 Treatment Arm vs Placebo Treatment Arm; Mean Change from Baseline in KDQOL-PFD: TRC101-Placebo; Test type: Superiority; p < 0.0001, ANCOVA — p-value based on analysis of covariance model with rank of change from baseline in total score as dependent variable; treatment (PBO or TRC101) as a fixed effect; and baseline total score, Baseline eGFR, Baseline Bicarbonate as continuous covariates

5. Secondary Outcome: Change From Baseline in the Duration of Repeated Chair Stand Test at the End of Treatment
Description: Change from baseline in the duration of repeated chair stand test at the end of treatment (Week 52). The five-times repeated chair stand test was used as a measure of lower extremity muscle strength. In this test, the time it took for a subject to repeatedly stand from a chair five times was recorded. This test is among the group of measures (gait speed, chair stand, and balance tests) comprising the Short Physical Performance Battery (SPPB), which has been used as a predictive tool for possible disability and for monitoring physical functioning in older people.
Time Frame: Baseline in the parent study, TRCA-301, to the Week 52 Visit in the extension study, TRCA-301E.
Population: as for outcome 2
Measure: Mean (Standard Error); unit: seconds
Arm/Group | TRC101 Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 112 | 77
seconds | -4.28 (1.240) | -1.42 (1.248)
Statistical Analysis 1: Comparison: TRC101 Treatment Arm vs Placebo Treatment Arm; Change from Baseline for Repeated Chair Stand Test: TRC101-Placebo; Test type: Superiority; p < 0.0001, ANCOVA

ADVERSE EVENTS:
Time Frame: Week 12 visit in the parent study, TRCA-301, to the Week 54 follow-up visit in the extension study, TRCA-301E.
Description: The TRCA-301E Safety Analysis Set included all subjects who received any amount of study drug (TRC101 or placebo) in TRCA-301E. Three subjects were excluded (2 TRC101, 1 placebo) because they entered TRCA-301E on a dose hold and remained on the dose hold for the duration of the study because their bicarbonate levels remained within the normal range.
Arm/Group | TRC101 Treatment Arm | Placebo Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/112 | 2/81
Serious Adverse Events (participants affected / at risk) | 2/112 | 4/81
Other Adverse Events (participants affected / at risk) | 78/112 | 39/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC101 Treatment Arm (N=112) | Placebo Treatment Arm (N=81)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC101 Treatment Arm (N=112) | Placebo Treatment Arm (N=81)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Headache (Nervous system disorders) | 17 (19) | 20 (22)
Flatulence (Gastrointestinal disorders) | 8 (8) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 5 (5)
Renal impairment (Renal and urinary disorders) | 5 (5) | 7 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 16 (19) | 8 (9)
Influenza (Infections and infestations) | 12 (13) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT03390842/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT03390842/SAP_001.pdf